CLINICAL TRIAL: NCT00369811
Title: Comparative Study of Oxycodone and Fentanyl Given Intravenously in the Treatment of Early Postoperative Pain After Laparoscopic Cholecystectomy
Brief Title: Oxycodone vs Fentanyl for Pain Treatment After Laparoscopic Cholecystectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Danish Pain Research Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OXFEN2006
Record Dates: First submitted 2006-08-28; First posted 2006-08-29 (Estimated); Last update posted 2007-11-19 (Estimated); Status verified 2007-11

CONDITIONS: Pain
Keywords: Cholecystectomy, postoperative
MeSH Terms: conditions — Pain | interventions — Oxycodone; Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Oxycodone, fentanyl

SUMMARY:
To evaluate the analgesic efficacy of oxycodone and fentanyl in the treatment of postoperative pain after laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* Planned outpatient laparoscopic cholecystectomy
* >18 years

Exclusion Criteria:

* Intolerance to study drugs
* Treatment with MAO inhibitors

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2006-08; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Pain intensity

CONTACTS AND LOCATIONS:
Overall Officials: Lone Nikolajsen, MD, PhD, Principal Investigator — Danish Pain Research Center, Aarhus University Hospital
Locations (1):
- Department of Anesthesiology, Aarhus University Hospital, Aarhus, Denmark